CLINICAL TRIAL: NCT00660348
Title: A Randomized Study of Optimal Pain Management: Standard Pain Control Versus Early Intervention With Intrathecal Therapy in Patients With Advanced Pancreatic Cancer
Brief Title: Standard Pain Control or Intrathecal Therapy in Controlling Pain in Patients With Locally Advanced, Unresectable, or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JHOC-J0724 CDR0000593173; P30CA006973 (NIH); JHOC-J0724; JHOC_NA_00009208
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Pain; Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas; pain; stage II pancreatic cancer
MeSH Terms: conditions — Pain; Pancreatic Neoplasms | interventions — Morphine

ARMS (2):
- morphine (Active Comparator): morphine given traditionally (IV, pill, patch). This is standard of care dosing.
  Interventions: Drug: morphine sulfate
- Intrathecal pump (Active Comparator): Pump internal used to deliver morphine. This is a newer method for delivery of morphine. Morphine is FDA approved for intrathecal use. The intrathecal pump will be titrated gradually to effect by the interventional pain medicine team. These are the maximum doses and concentrations in keeping with the Polyanalgesic Consensus Conference guidelines: Dose (mg/day):15 ; Conc (mg/cc): 20
  Interventions: Device: Medtronic intrathecal pump

INTERVENTIONS:
Drug: morphine sulfate — This is morphine given in the traditional methods.
  Arms: morphine
Device: Medtronic intrathecal pump — This pump will be inserted into the research subject and then the pump will deliver morphine.
  Arms: Intrathecal pump

SUMMARY:
RATIONALE: Giving medications in different ways may change their effectiveness in controlling pain. It is not yet known whether intrathecal therapy is more effective than standard therapy in controlling pain in patients with pancreatic cancer.

PURPOSE: This randomized clinical trial is studying standard pain control to see how well it works compared with intrathecal therapy in controlling pain in patients with locally advanced, unresectable, or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the effectiveness of pain control comprising intrathecal opioid delivery versus the standard analgesia-delivery method in patients with locally advanced, unresectable, or metastatic pancreatic cancer.

Secondary

* To assess the difference of a total amount of opioid consumption (parenteral morphine equivalent) between two different opioids-delivery groups at one month of treatment.
* To assess the average of percent change in Karnofsky performance status with respect to the baseline status between two different analgesic-delivery groups at one month of treatment.
* To assess the difference in quality of life between two different opioids-delivery groups at one month of treatment using the EORTC QLQ-C30.
* To assess overall survival of these patients.
* To assess the safety profile of two different analgesic-delivery methods (i.e., adverse event and serious adverse event).

OUTLINE: Patients are stratified according to Karnofsky performance status (60-80% vs > 80%). Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard pain management): Patients are evaluated by the JHH Pain Medicine Integrated Team for pain, for the potential of diagnostic/neurolytic celiac plexus block, and undergo the institution of or modification of or continuation and titration of oral or parenteral analgesics. Patients undergo a limited, problem-oriented physical exam including weight, vital signs, Karnofsky performance status (KPS), assessment of previously abnormal findings or new complaints, pain scores, analgesia consumption, side effects (i.e., sleepiness, nausea, pruritus, and constipation), and quality-of-life score (EORTC QLQ-C30) once every 2 weeks for 3 months and then once a month thereafter. Patients also keep a diary of pain scores and side effects during the trial. Patients may have their treatment titrated as needed to control their pain. Patients who are not adequately pain controlled or develop debilitating side effects from their therapy may be managed by adjuvant analgesics or be allowed to crossover into the treatment arm of the study to provide compassionate care.
* Arm II (intrathecal therapy): Patients undergo implantation of a Medtronic intrathecal pump and catheter system for delivery of morphine sulfate directly into the spinal fluid. Following implantation, patients undergo a limited, problem-oriented physical exam including vital signs, KPS, assessment of previously abnormal findings or new complaints, pain scores, analgesia consumption, and quality-of life-score (EORTC QLQ-C30) once every 2 weeks for 3 months and then once a month thereafter. Patients are also evaluated by the Interventional Pain Treatment Team for wound status, presence of symptoms of post-dural puncture headache, signs of infection, or meningitis. Patients are followed by the JHH Pain Medicine Integrated Team for evaluation of pain and for institution of or modification of or continuation and titration of oral or parenteral analgesics.

After completion of study treatment, patients are followed for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed adenocarcinoma of the pancreas

  * Mixed adenocarcinoma tumors allowed provided the predominant invasive component of the tumor is adenocarcinoma
* Locally advanced, unresectable, or metastatic disease
* Patients must be within two months of diagnosis or have started chemotherapy within 60 days of study
* Average pain score ≥ 4/10 over a 7-day period on a verbal numerical rating scale

Exclusion criteria:

* Known brain metastases
* Tumor with clinically significant obstruction of the spinal canal

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* ANC ≥ 1,500 cells/mm³
* Hematocrit ≥ 28%
* WBC ≥ 3,500 cells/mm³
* Platelets ≥ 90,000/mm³
* Serum creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.5 mg/dL
* AST/ALT ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* INR ≤ 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Mini-mental status exam score ≥ 22

Exclusion criteria:

* Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this therapy, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Active peptic ulcer disease
* Active infections
* Insensitive to opioid medication for cancer pain
* Insufficient tissue or decubitus ulcer near device implantation site
* Current history of substance abuse

PRIOR CONCURRENT THERAPY:

* Minor procedures (i.e., dental work or skin biopsy), tumor biopsies, and biliary stent placement are allowed
* No prior surgical procedures affecting absorption
* Prior or other concurrent pain medications are allowed
* Concurrent chemotherapy or radiotherapy allowed at the discretion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Erdek, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine: morphine given traditionally (IV, pill, patch)
  morphine sulfate: This is morphine given in the traditional methods.
- Intrathecal Pump: Pump internal used to deliver morphine. This is a newer method for delivery of morphine.
  Medtronic intrathecal pump: This pump will be inserted into the research subject and then the pump will deliver morphine.
Period: Overall Study
Arm/Group | Morphine | Intrathecal Pump
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Intrathecal Pump | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] — Years
  years | 55 [55 to 55] |  | 55 [55 to 55]
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Per Arm With Decrease in Pain Scores
Description: The primary objective of this study is to compare the effectiveness of pain control between intrathecal opioid delivery and standard analgesia delivery method in patients with locally advanced unresectable or metastatic pancreatic cancer. The primary end point is the number of subjects on each arm showing a decrease in the change in VAS self-assessment pain intensity rating (VAS pain rating) at one month from initial treatment with respect to the baseline pain score. The change is defined as (the Pain Score at one month of the treatment - the Pain Score at baseline). Serial pain scores will be collected at all assessment time points. Min: zero cm. Max 10cm. A higher value means worse pain. Subjects on each arm will report pain on a 10 cm Visual Analogue Scale (VAS) pain rating scale, by making a mark on the 10cm horizontal line with a pen and study team will measure distance from the mark to the start of the scale, which will indicate pain score (eg 1 cm, 3 cm 6 cm, etc.).
Time Frame: 1 month
Population: One subject was enrolled, and baseline pain score was obtained on questionnaire, but the subject came off-study before follow-up pain score could be collected. Study terminated shortly thereafter. No outcome data were collected.
Arm/Group | Morphine | Intrathecal Pump
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Morphine | Intrathecal Pump
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=1) | Intrathecal Pump (N=0)
epigastric pain (upper quadrant) (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3 epigastric pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=1) | Intrathecal Pump (N=0)
reflux intermittent (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 1
fatigue (General disorders) | 1 (1) | 0 (0) — grade 1

LIMITATIONS AND CAVEATS:
Subject started study 7/14/2010, but withdrew her consent on 7/24/2010 due to increased upper quadrant pain. One subject enrolled. She withdrew consent before study team could collect any follow-up data. We do not have any participants to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes